CLINICAL TRIAL: NCT01963741
Title: Leukotriene D4 Nasal Provocation Test: Rationale, Methodology, Diagnostic Value and Its Impact on Airway Inflammation in Allergic Rhinitis With or Without Asthma
Brief Title: Leukotriene D4 Nasal Provocation Test in Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jinping Zheng, Professor,Guangzhou institute of respiratory disease, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: LTD4NAPT201218
Record Dates: First submitted 2013-08-27; First posted 2013-10-16 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: Leukotriene D4; allergic rhinitis; nasal airway resistance; nasal provocation test; nasal hyperreactivity; airway inflammation; asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma | interventions — Leukotriene D4; Histamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- leukotriene D4 (Experimental): Nasal provocation test was induced by leukotriene D4 with a stepwisely concentration method (4 mcg/ml, 8 mcg/ml, 16 mcg/ml).
  Interventions: Drug: histamine
- histamine (Experimental): Nasal provocation test was induced by histamine with a stepwisely concentration method (0.4 mg/ml, 0.8 mg/ml, 1.6 mg/ml, 3.2mg/ml).
  Interventions: Drug: leukotriene D4

INTERVENTIONS:
Drug: leukotriene D4 — Nasal challenge using 16% ethanol diluent, the concentration of which corresponded to the highest concentration of LTD4, was undertaken for exclusion of subjects hypersensitive to ethanol or saline. The LTD4 challenge could be initiated provided that NAR increase was <30%. Ranges of 4 to 16 mcg.mL-1 LTD4 diluents were applied for a double-fold increment approach at intervals of 6 minutes.
  Other Names: Cayman chemical company (1-800-364-9897 Cat 20310).
  Arms: histamine
Drug: histamine — Nasal challenge using 0.9% saline, was undertaken for exclusion of subjects hypersensitive to saline. The histamine nasal challenge could be initiated provided that NAR increase was <30%. Ranges of 0.4 to 3.2 mg.mL-1 histamine diluents were applied for a double-fold increment approach at intervals of 3 minutes.
  Other Names: Guangzhou chemical company (serial number: 1703 )
  Arms: leukotriene D4

SUMMARY:
Leukotrienes play critical roles in the inflammatory process in allergic rhinitis and bronchial asthma, therefore, anti-leukotriene therapy is part of treatment for asthma. However, not all allergic rhinitis accompanied with or without asthma treated with anti-leukotriene were effective. So it is critical to develop a method to identify the response subgroup. In this study, it is assumed that nasal physiological responsiveness to leukotriene nasal provocation test (NPT) is able to gain evidence on the effect of leukotriene on the development of allergic rhinitis and asthma, and is helpful to the use of anti-leukotriene agent. The purpose of the study is to establish the methodology and diagnostic value of leukotriene D4 (LTD4) nasal provocation.

DETAILED DESCRIPTION:
Nasal provocation test induced by LTD4 will be conducted by measuring nasal airway resistance and airway symptoms in a stepwise concentration of LTD4 by nasal spray. Inflammation biomarkers, such as eosinophilic granulocyte in sputum and nasal lavage, fractional exhaled nitric oxide(FeNO), and lung function before and after nasal provocation will be studied to explore the impact of LTD4 nasal provocation test on airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with allergic rhinitis accompanied with or without asthma
* positive skin prick test (SPT)
* had no acute upper or lower airway infection 2 weeks prior to study
* no oral or nasal anti-histamines
* no leukotriene receptor antagonists for 1 week
* no oral or nasal and inhaled corticosteroids for 2 weeks

Exclusion Criteria:

* smokers
* a past confirmed history of chronic respiratory disease other than asthma
* other severe systemic diseases (myocardial infarction, malignant tumor, etc.)
* under immunotherapy
* unable to complete the test or had limited understanding
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants positive response to leukotriene D4 or histamine nasal provocation test | Until 1 hour after the nasal provocation test
  Nasal airway resistance measured by positive anterior rhinomanometry. Concentration induced 60% increase of nasal airway resistance (PC60-NAR) will be measured and reported; Composite symptoms score defined by reichmann H and his colleagues showed as follows:3-5 sneezes = 1 point (pt), >5 sneezes = 2 points (pts); rhinorrhoea < 1 milliliter (mL) = 1 pt, rhinorrhoea > 1 milliliter = 2 pts; pruritus of the palate or ear or eye= 1 pt, conjunctivitis or cough or urticaria or difficult breathing= 2 pts. Total score ranges from 0 to 6 pts. Positive response to LTD4 nasal provocation test was defined as PC60-NAR less than 16mcg/mL or the symptom score higher than 3.

SECONDARY OUTCOMES:
Change from baseline of eosinophils in sputum and nasal lavage and fractional exhaled nitric oxide (FeNO) | 4 and 24 hours after the nasal provocation test
  Biomarkers in upper and lower airways such as eosinophils in sputum and nasal lavage and fractional exhaled nitric oxide (FeNO) will be studied.

OTHER OUTCOMES:
Change from baseline of cumulative dosage of methacholine causing a 20% fall in forced expiratory volume in 1 second (PD20FEV1-MCH) | Half an hour after nasal provocation test
  The increase of brochial hyperresponsiveness induced by nasal provocation test was assessed by the decrease of cumulative dosage of methacholine causing a 20% fall in forced expiratory volume in 1 second (PD20FEV1-MCH).
Peak Nasal Inspiratory Flow (PNIF) | 3 minutes after each concentration of provocation agent administrated into the nostrils
  The peak nasal inspiratory flow (PNIF) is measured by PNIF meter (in-check dial, Clement Clarke International Ltd.); Change from baseline of peak nasal inspiratory flow (PNIF) at the end of nasal provocation test will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, professor, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Busse WW. The role of leukotrienes in asthma and allergic rhinitis. Clin Exp Allergy. 1996 Aug;26(8):868-79. PMID 9011329
- [Background] Howarth PH, Salagean M, Dokic D. Allergic rhinitis: not purely a histamine-related disease. Allergy. 2000;55 Suppl 64:7-16. doi: 10.1034/j.1398-9995.2000.00802.x. PMID 11291780
- [Background] Patel P, Philip G, Yang W, Call R, Horak F, LaForce C, Gilles L, Garrett GC, Dass SB, Knorr BA, Reiss TF. Randomized, double-blind, placebo-controlled study of montelukast for treating perennial allergic rhinitis. Ann Allergy Asthma Immunol. 2005 Dec;95(6):551-7. doi: 10.1016/S1081-1206(10)61018-6. PMID 16400895
- [Background] Philip G, Williams-Herman D, Patel P, Weinstein SF, Alon A, Gilles L, Tozzi CA, Dass SB, Reiss TF. Efficacy of montelukast for treating perennial allergic rhinitis. Allergy Asthma Proc. 2007 May-Jun;28(3):296-304. doi: 10.2500/aap.2007.28.3000. PMID 17619558
- [Background] Price DB, Swern A, Tozzi CA, Philip G, Polos P. Effect of montelukast on lung function in asthma patients with allergic rhinitis: analysis from the COMPACT trial. Allergy. 2006 Jun;61(6):737-42. doi: 10.1111/j.1398-9995.2006.01007.x. PMID 16677244
- [Background] Pinar E, Eryigit O, Oncel S, Calli C, Yilmaz O, Yuksel H. Efficacy of nasal corticosteroids alone or combined with antihistamines or montelukast in treatment of allergic rhinitis. Auris Nasus Larynx. 2008 Mar;35(1):61-6. doi: 10.1016/j.anl.2007.06.004. Epub 2007 Sep 7. PMID 17826020
- [Background] Nayak A, Langdon RB. Montelukast in the treatment of allergic rhinitis: an evidence-based review. Drugs. 2007;67(6):887-901. doi: 10.2165/00003495-200767060-00005. PMID 17428106
- [Background] Virchow JC, Bachert C. Efficacy and safety of montelukast in adults with asthma and allergic rhinitis. Respir Med. 2006 Nov;100(11):1952-9. doi: 10.1016/j.rmed.2006.02.026. Epub 2006 Apr 12. PMID 16626955
- [Background] Bisgaard H, Olsson P, Bende M. Effect of leukotriene D4 on nasal mucosal blood flow, nasal airway resistance and nasal secretion in humans. Clin Allergy. 1986 Jul;16(4):289-97. doi: 10.1111/j.1365-2222.1986.tb01960.x. PMID 2427255
- [Background] Miadonna A, Tedeschi A, Leggieri E, Lorini M, Folco G, Sala A, Qualizza R, Froldi M, Zanussi C. Behavior and clinical relevance of histamine and leukotrienes C4 and B4 in grass pollen-induced rhinitis. Am Rev Respir Dis. 1987 Aug;136(2):357-62. doi: 10.1164/ajrccm/136.2.357. PMID 3039881
- [Background] Brozek JL, Baena-Cagnani CE, Bonini S, Canonica GW, Rasi G, van Wijk RG, Zuberbier T, Guyatt G, Bousquet J, Schunemann HJ. Methodology for development of the Allergic Rhinitis and its Impact on Asthma guideline 2008 update. Allergy. 2008 Jan;63(1):38-46. doi: 10.1111/j.1398-9995.2007.01560.x. PMID 18053015
- [Background] Riechelmann H, Bachert C, Goldschmidt O, Hauswald B, Klimek L, Schlenter WW, Tasman AJ, Wagenmann M; German Society for Allergology and Clinical Immunology (ENT Section); Working Team for Clinical Immunology. [Application of the nasal provocation test on diseases of the upper airways. Position paper of the German Society for Allergology and Clinical Immunology (ENT Section) in cooperation with the Working Team for Clinical Immunology]. Laryngorhinootologie. 2003 Mar;82(3):183-8. doi: 10.1055/s-2003-38411. No abstract available. German. PMID 12673517
- [Background] Guan W, Zheng J, Gao Y, Jiang C, Xie Y, An J, Yu X, Liu W, Zhong N. Leukotriene D4 and methacholine bronchial provocation tests for identifying leukotriene-responsiveness subtypes. J Allergy Clin Immunol. 2013 Feb;131(2):332-8.e1-4. doi: 10.1016/j.jaci.2012.08.020. Epub 2012 Oct 4. PMID 23040886
- [Background] Guan W, Zheng J, Gao Y, Jiang C, An J, Yu X, Liu W. Leukotriene D4 bronchial provocation test: methodology and diagnostic value. Curr Med Res Opin. 2012 May;28(5):797-803. doi: 10.1185/03007995.2012.678936. Epub 2012 May 3. PMID 22435894
- [Derived] Zhu Z, Xie Y, Guan W, Gao YI, Xia S, Liang J, Zheng J. Leukotriene D4 nasal provocation test: Rationale, methodology and diagnostic value. Exp Ther Med. 2016 Jul;12(1):525-529. doi: 10.3892/etm.2016.3324. Epub 2016 May 10. PMID 27347089